CLINICAL TRIAL: NCT04693130
Title: Effects of Mindfulness-based Prenatal Education on Biopsychological Health for Prenatal Mental Disorders Women
Brief Title: Mindfulness-based Prenatal Education on Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taipei University of Nursing and Health Sciences (Other)
Responsible Party: Principal Investigator, Wan-Lin Pan, Nursing department, National Taipei University of Nursing and Health Sciences
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 108-E-14
Record Dates: First submitted 2020-12-24; First posted 2021-01-05 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Depression, Anxiety
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness-based prenatal education (Experimental): The intervention includes 3-hour classes per week during the duration of eight weeks and a 7- hour silent meditation practice as well.
  Interventions: Behavioral: Mindfulness-based prenatal education
- Hospital-based antenatal education (Placebo Comparator): Hospital-based antenatal education program.
  Interventions: Behavioral: Hospital-based antenatal care

INTERVENTIONS:
Behavioral: Mindfulness-based prenatal education — Mindfulness-based prenatal education involves mindfulness breathing and other skills with mindfulness meditations.
  Arms: Mindfulness-based prenatal education
Behavioral: Hospital-based antenatal care — Hospital-based antenatal care involves all aspects of pregnancy, childbirth and postpartum.
  Arms: Hospital-based antenatal education

SUMMARY:
The purpose of this study is to explore the differences between stress, anxiety, depression, mindfulness, mother and infants bonding, salivary amylase activity, and postnatal maternal outcomes for prenatal mental disorders in women with mindfulness prenatal education program

DETAILED DESCRIPTION:
The aim of this study was to test the efficacy of a Mindfulness prenatal education program in reducing pregnant women's perceived stress, anxiety, depression, mindfulness, mother and infant bonding, and salivary alpha-amylase compared to a control group. The investigators hypothesize that using the mindfulness prenatal education program by the study group will lead to improved related mood symptoms compared with the control group.

Randomized Controlled Trial comparing two education programs with health and singleton pregnant women is run by the Random Allocation Software (Saghaei, 2004). Use the G-Power 3.1.9 windows: repeated measures and between factors among two groups to calculate the number of samples, and setting the power = .8, α = .05, effect size = .25. The estimated number of samples may be lost 30%, total 102 samples.

ELIGIBILITY:
Inclusion Criteria:

* Subjects were at the age over 20
* Could speak and read Chinese fluently
* Willing and be ale to attend the education program

Exclusion Criteria:

* Taking medication for diagnosing mental illness
* With complicated or high-risk pregnancies

Min Age: 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2020-12-24 (Actual); Primary Completion 2022-03-03 (Actual); Study Completion 2023-02-03 (Actual)

PRIMARY OUTCOMES:
stress | baseline , and at eight weeks (after the intervention), 36 weeks of gestation, and the follow-up at 2 , 4 months postpartum
  Perceived stress scale, that was 10 items to determine the self-perceived levels of unpredictability, lack of control, and burden during the last month of pregnancy. Responses are rated from 0 (never) to 4 (very often), with higher scores corresponding to higher perceived stress

SECONDARY OUTCOMES:
depression | baseline , and at eight weeks (after the intervention), 36 weeks of gestation, and the follow-up at 2 , 4 months postpartum
  Edinburgh Perinatal Depression Scale, that was 10-question questionnaire provides a valuable and efficient way to identify patients at risk of perinatal depression. Each item is scored from 0 to 3, with item scores summed to produce a total score

OTHER OUTCOMES:
mindfulness | baseline , and at eight weeks (after the intervention), 36 weeks of gestation, and the follow-up at 2 , 4 months postpartum
  The Five Facet Mindfulness Questionnaire, that was 39-item is based on factor analysis. The five facets of the FFMQ include: observing, describing, acting with awareness, non-judging of inner experience, and non-reactivity to inner experience. Scoring uses a 5-point Likert scale, with 1 representing "never or very rarely true" and 5 representing "very often or always true"
anxiety | baseline , and at eight weeks (after the intervention), 36 weeks of gestation.
  The Pregnancy-Related Thoughts Questionnaire (PRT), which uses a 10-item scale to measure a person's attention to baby health, labor, childbirth, and caring for babies over the past 7 days.indicated population by Robles et al. It consists of 21 items that evaluate symptoms of anxiety on a four-point Likert scale ranging from 0 = "not at all" to 3 = "severely." The anxiety level was scored using ordinal categories: minimal (1-5 points), mild (6-15), moderate (16-30) and severe (31-63)
bonding | the follow-up at 2 , 4 months postpartum.
  The mother's feelings or attitudes toward her baby were assessed using the Postpartum Bonding Questionnaire (PBQ).

CONTACTS AND LOCATIONS:
Overall Officials: Wan-Lin Pan, PHD, Principal Investigator — National Taipei University of Nursing and Health Sciences
Locations (1):
- Wan-Lin Pan, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pan WL, Lin LC, Kuo LY, Chiu MJ, Ling PY. Effects of a prenatal mindfulness program on longitudinal changes in stress, anxiety, depression, and mother-infant bonding of women with a tendency to perinatal mood and anxiety disorder: a randomized controlled trial. BMC Pregnancy Childbirth. 2023 Jul 31;23(1):547. doi: 10.1186/s12884-023-05873-2. PMID 37525110